CLINICAL TRIAL: NCT04240028
Title: The Cognitive-Prefrail Syndrome and Its Association With Adverse Health Outcomes: Results From the NuAge Observational Population-based Study
Brief Title: The Cognitive-Prefrail Syndrome and Its Association With Adverse Health Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Professor of Geriatrics, Holder of the Dr. Joseph Kaufmann Chair in Geriatric Medicine, Clinician Scientist, Director of Centre of Excellence on Longevity, Jewish General Hospital
Other Study IDs: 2020-2029
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Cognitive-prefrailty; Prefrailty; Motoric Cognitive Risk Syndrome
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with prefrailty: This is defined as a co-existing prefrailty using the Fried criteria. Frailty defined by the CHS index as proposed by Fried et al. will be identified by the presence of ≥ 3 of the following 5 components: 1) Shrinking as identified by an unintentional weight loss of ≥ 5% between two assessments, 2) Weakness as identified by a maximal grip strength in the lowest quintile stratified by body mass index quartile; 3) Poor energy as identified by an answer of "no" to the question "Do you feel full of energy?" from the 30-item Geriatric Depression Scale; 4) Slowness as identified by an average walk speed in the lowest quintile stratified by median standing height, and 5) Low physical activity level as identified by a PASE score in the lowest quintile. Participants with none of the above components will be considered to be vigorous and those with 1 or 2 components will be considered to be in a prefrail stage.
  Interventions: Other: Data Collection
- Individuals with cognitive-prefrailty: A combination of prefrailty stage using Fried criteria and subjective cognitive impairment (SCI).
  The IANA/IAGG consensus defines cognitive frailty as CDR = 0.5 and frailty by the Fried criteria.SCI will be defined using a proxy for subjective cognitive complaint (i.e. memory complaint) and following the procedure used in previous multicenter prevalence studies on MCR syndrome. Memory complaint used to define MCR syndrome was based on standardized memory loss question on the 15-item or 30-item Geriatric Depression Scale (GDS; "Do you feel you have more problems with memory than most?"). Memory complaint in our study will be elicited from this item of 30-item GDS.
  Interventions: Other: Data Collection
- Individuals with MCR: The diagnosis of MCR syndrome will be made following the criteria of Verghese et al. 5: a combination of subjective cognitive complaint, in particular of memory complaint, with the presence of an objective slow gait and the absence of dementia or mobility disability. MCR syndrome will be defined at baseline assessment and each year of follow-up period. Slow gait speed will be defined as gait speed that is one standard deviation (SD) or more below age-and sex-appropriate mean values established in the present cohort like in previous studies. The mean value and SD of female and male will be determined separately. Gait speed was determined from the 3-meter walking test using the best time of the two trials recorded and expressed as meters per second.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — The NuAge study has been designed to investigate nutrition as a determinant of successful aging in older men and women in Quebec. This study is based on a population-based observational cohort design that initially recruited healthy community-dwellers with age ranged from 67 to 82 years (51.8% women) between January 2004 and April 2005. All participants lived in the areas of Montreal, Laval, and Sherbrooke in the Province of Quebec, Canada. After recruitment, they have been followed for 3 years with one clinical follow-up assessment each year (i.e.; 4 data collection time). A previous analysis performed on the NuAge study database has shown a significant decline of physical and cognitive performances with time (respectively an average of 10% and 2%), participants with lower physical performance showing lower cognitive performance.

SUMMARY:
Lay Summary Older adults who are prefrail (an intermediate, potentially reversible stage between robustness and frailty) with early symptoms of cognitive impairment are a segment of the population that have hitherto remained "silent" and are currently not targets for screening and intervention. These individuals require early identification for preventive interventions to reduce disability, dependency and improve quality of life. To date, there is still no accepted definition of individuals upstream in the spectrum of physical frailty and cognitive impairment. Determining the prevalence and predictive ability of various definitions of co-existent frailty and cognitive impairment could identify older adults at greatest risk of adverse health outcomes. Therefore, the researchers aim to examine and compare (1) the prevalence of cognitive-prefrailty, prefrailty (IANA/IAGG consensus definition) and MCR syndromes, (2) the incidence and predictive ability of these three syndromes for adverse health outcomes including cognitive impairment and decline, dementia, physical functional impairment and decline, falls, hospitalization and mortality in older Quebec community dwellers.

DETAILED DESCRIPTION:
Scientific Summary

Background Cognitive frailty is the simultaneous presence of both physical frailty and cognitive impairment, excluding concurrent dementia. This condition confers a greater risk of incident cognitive impairment and decline, dementia, falls and disabilities compared to either condition alone. Current definitions of co-existent frailty and cognitive impairment exist, including the International Academy on Nutrition and Aging (IANA) and the International Association of Gerontology and Geriatrics (IAGG) consensus for cognitive frailty. There is also an analogous construct known as the motoric cognitive risk syndrome (MCR) associating slow gait speed and subjective cognitive impairment (SCI). Current operational criteria identify individuals later in the trajectory of frailty and cognitive decline, which may be too late for effective interventions. The researchers propose to define a new and early condition in the spectrum of Cognitive frailty known as "cognitive-prefrailty", which is a combination of prefrailty stage and SCI.

Overall objective This study aims to determine and compare (1) the prevalence of cognitive-prefrailty, cognitive frailty (IANA/IAGG consensus definition) and MCR syndromes, (2) the incidence and predictive ability of these three syndromes for adverse health outcomes including cognitive impairment and decline, dementia, physical functional impairment and decline, falls, hospitalization and mortality in older community dwellers.

Methods This study will use the database of the "Nutrition as a determinant of successful aging: The Quebec longitudinal study" (NuAge) study, which is a population-based observational cohort hat recruited healthy community-dwellers with age ranged from 67 to 84 years (51.8% women) between November 2003 and June 2005, and followed them during 4 years. Cognitive-prefrailty, prefrailty and MCR will be defined using information collected at the baseline assessment. Incident adverse health outcomes including cognitive impairment and decline, dementia, physical functional impairment and decline, falls, hospitalization and mortality have been recorded during the 4-years follow-up period.

Anticipated results Prefrailty (an intermediate and potentially reversible stage between robust and frailty) and SCI occur upstream in the continuum of frailty and cognitive decline and hence constitute more suitable targets for screening and early intervention in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Be participants of the NuAge study who agreed to be part of the NuAge Database and Biobank for future research purposes

Exclusion Criteria:

* Missing data at baseline and follow-up assessments
* Participants' refusal to use their data for a purpose not identified during their recruitment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Individuals eligible for this study will be participants of the NuAge study (n=1,793). All included participants of NuAge Study were healthy and, in particular, they were cognitively intact at baseline and had no mobility disability.
Sampling Method: Non-Probability Sample
Enrollment: 1741 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment | 1 day
  Cognitive status has been measured using the Modified Mini-Mental State (3MS)17 in the NuAge study. The 3MS test has a score range of 1-100. Baseline value and change over the three years of follow-up will be used. Cognitive impairment will be considered when 3MS score < 79.
Cognitive decline | 1 day
  From T2 to T4 annual variation of 3MS score expressed in percentage between T1-T2, T2-T3 and T3-T4 will be calculated using the formula: ((3MS Tn+1 - 3MS Tn+1) / ((3MS Tn+1 + 3MS Tn+1) / 2)) x 100.
Incident dementia | 1 day
  From T2 to T4, incident dementia will be considered if 3MS score is ≤79/100 and simplified instrumental activity daily living score is <4
Physical functional impairment | 1 day
  A sex-specific global measure of physical performance will be computed as the sum of scores in four tests: standing balance, walking speed (normal and fast), chair stands, and timed "Up & Go" according to a slightly modified method proposed by Guralnik and colleagues.18 The validity of this global measure has been previously reported in this population.19 Four levels of physical performance will be created for each of the five tests. A score from 1 (slowest) to 4 (fastest) is assigned according to the quartile of time needed to carry out the test. With the exception of standing balance, the lowest quartile indicates the best (shorter duration) score. The reverse is true with respect to standing balance. A score of 0 was assigned to those who could not do or did not complete the test because they felt unable to do so. Possible scores range from 0 (worst) to 20 (best).
Physical functional Decline | 1 day
  From T2 to T4 annual variation of Physical functional score expressed in percentage between T1-T2, T2-T3 and T3-T4 were calculated using the formula: ((score Tn+1 - score Tn+1) / ((score Tn+1 + score Tn+1) / 2)) x 100
Falls | 1 day
  number of falls
Hospitalizations | 1 day
  Number of hospitalization
Mortality | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — McGill University, Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada